CLINICAL TRIAL: NCT02999620
Title: A Single Center, Randomized, Double-blind, Placebo Controlled, Two-way Crossover Study to Determine the Fat Losses in Stool Associated With Alpha-CD Use as Compared to Placebo Using a Radiotracer
Brief Title: FBCx (Alpha-CD) Mechanism of Action Trial
Acronym: FMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SFI Research (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SFIR-FMAT-US01
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha-cycoldextrin (Active Comparator): All subjects randomized to receive Alpha-cycoldextrin will orally ingest two tablets containing Alpha-cyclodextrin, with their standardized liquid breakfast (100 micro Ci of [3H]triolein and 20 micro Ci of [14C]tripalmitin). The tablets will be consumed with 150 ml of still water immediately prior to consuming each meal. Subjects will be observed for a period of 48 hours as an in-patient, and then an additional 24 hours as an out-patient. During this time they will undergo a meal fatty acid metabolism study, through blood and fecal sampling, to assess meal fatty acid oxidation and storage.
  Interventions: Dietary Supplement: Alpha-cyclodextrin
- Placebo (Placebo Comparator): All subjects randomized to receive placebo will orally ingest two placebo tablets with their standardized liquid breakfast (100 micro Ci of [3H]triolein and 20 micro Ci of [14C]tripalmitin). The tablets will be consumed with 150 ml of still water immediately prior to consuming each meal. Subjects will be observed for a period of 48 hours as an in-patient, and then an additional 24 hours as an out-patient. During this time they will undergo a meal fatty acid metabolism study, through blood and fecal sampling, to assess meal fatty acid oxidation and storage.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-cyclodextrin — Alpha-cyclodextrin (α-CD) is a soluble dietary fiber that has a history of use in foods and as a pharmaceutical excipient. Recently the ability of the fiber to bind to dietary fat has led to further investigation of the possible health benefits of dietary supplementation with this fiber.
  Other Names: Calorease, Nuvexa, Mirafit, FBCx, Alfadex
  Arms: Alpha-cycoldextrin
Dietary Supplement: Placebo — Identical looking placebo tablet to active (Alpha-cyclodextrin)
  Arms: Placebo

SUMMARY:
To determine the fat losses in stool associated with alpha-CD use in healthy volunteers, as compared to placebo when consumed with a standardized radiolabeled fatty meal.

DETAILED DESCRIPTION:
This clinical investigation will determine the fat losses in stool associated with alpha-CD use as compared to placebo when ingested with a standardized liquid breakfast (100 microCi of [3H]triolein) and 20 microCi of [14C]tripalmitin). The ingested dose will be 2 g of α-CD at each of three meals per day for 2 days.

Eight subjects will be recruited in a two-way crossover design consisting of two treatment periods.

Treatment 1 requires all subjects to receive α-CD and a meal containing the fatty acid radiotracers Treatment 2 requires all subjects to receive placebo and a meal containing the fatty acid radiotracers All subjects will be observed for 48 hours as an in-patient, and a further 24 hours as an out-patient following the meal containing the radiotracer and will then undergo at least a further ≥ 14 day washout period before crossing over to the alternate treatment.

All subjects randomized to the α-CD treatment arm will receive 2 g of α-CD (2 x 1 g tablets), at each of three meals per day for 2 days. During the placebo phase, all subjects will receive two identical-looking placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy weight stable individuals (defined as a BMI of ≥18.5 and <27, and stable for at least the preceding two months from Screening)
* Not pregnant, and if of childbearing potential, agrees to use adequate birth control (hormonal or barrier method of birth control or abstinence) prior to study entry and during the trial and agrees not to donate sperm or ova, for the duration of the study
* Subjects ≥ 18 - ≤60 years of age at screening
* Consistent regular bowel movement (defined as between 3 times a day to 1 time per day)
* Provide Informed Consent
* Willing and able to complete study procedures within the study timelines
* Adequate renal function: serum creatinine less than 1.5 x upper limit of normal (ULN)
* Adequate liver function: serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) and serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) ≤ 2 × ULN and serum bilirubin ≤ 1.5 × ULN unless Gilbert's syndrome has previously been confirmed for the subject
* Adequate bone marrow function: white blood cells (WBCs) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, hemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/mm3

Exclusion Criteria:

* Evidence of chronic pancreatitis
* Evidence of irritable bowel syndrome (medical or self-diagnosed)
* Previous gallbladder surgery
* Use of enemas and/or suppositories within 30 days of Screening
* Consuming ≥ 375 mg of caffeine per day (equivalent to 5 serves of 1 oz. restaurant style espresso per day)
* History of febrile illness within 5 days prior to Screening
* Evidence or history of substance or alcohol abuse
* History of major depression (per DSM4 criteria), bipolar disorder, or schizophrenia
* Current use of prescription or non-prescription weight loss products (≥ 2 week washout period is required to become eligible)
* Smoking ≥ 30 cigarettes (one pack) per week
* Significant dietary restrictions (incl. vegan, vegetarian diets and any subject not prepared to consume any of the standardized food/s
* Evidence of an active eating disorder (incl. anorexia nervosa, bulimia, and/or obsessive compulsive disorders)
* Use of other investigational agent(s) at the time of enrollment, or within 30 days or five half-lives of enrollment, whichever is longer
* Pregnant or lactating
* Current use of any medication known to affect gut motility
* History of malignancy, treated or untreated, within the past five years, with the exception of non-melanoma skin cancer and cervical carcinoma in situ
* A known history of hypersensitivity to any of the α-CD components
* Any other health condition that would preclude participation in the study in the judgment of the principal investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Radiolabeled lipid content in stool | 72 hours
  The primary endpoint for this investigation is to measure the total excretion of radiolabeled fat in feces over 72 hours.

SECONDARY OUTCOMES:
Blood glucose levels | 6 hours
  Blood Glucose will be measured hourly from fasting to 6 hours post radiotraced meal on the first day of each treatment period.

OTHER OUTCOMES:
Blood Trigliceride Levels | 6 hours
  Blood Triglyceride concentrations will be measured hourly from fasting to 6 hours post radiotraced meal on the first day of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Comerford KB, Artiss JD, Jen KL, Karakas SE. The beneficial effects of alpha-cyclodextrin on blood lipids and weight loss in healthy humans. Obesity (Silver Spring). 2011 Jun;19(6):1200-4. doi: 10.1038/oby.2010.280. Epub 2010 Dec 2. PMID 21127475
- [Result] Jarosz PA, Fletcher E, Elserafy E, Artiss JD, Jen KL. The effect of alpha-cyclodextrin on postprandial lipid and glycemic responses to a fat-containing meal. Metabolism. 2013 Oct;62(10):1443-7. doi: 10.1016/j.metabol.2013.05.015. Epub 2013 Jun 24. PMID 23806736